CLINICAL TRIAL: NCT04468165
Title: Effectiveness and Safety of Generic Delayed-Release Dimethyl Fumarate (Sclera® or Marovarex ®, Hikma) in Routine Medical Practice in the Treatment of Relapsing-Remitting Multiple Sclerosis in MENA Region
Status: Completed | Type: Observational
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HIK-DMF-2020-01
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Dimethyl Fumarate; Generic Dimethyl Fumarate; Delayed-Release Dimethyl Fumarate; Disease Modifying Treatments; Nervous System; Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis; Cohort Study; Observational Study; Effectiveness; Safety; Health Related Quality of life
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Neurologic Manifestations; Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dimethyl Fumarate (DMF) — Gastro-resistant Hard Capsules. Each capsule contains 240mg or 120mg Dimethyl Fumarate
  Other Names: Sclera ®, Hikma; Marovarex ®, Hikma

SUMMARY:
The purpose of this observational study is to evaluate the effectiveness, safety and health related quality of life of Generic DMF (Sclera® or Marovarex ®, Hikma) in patients undergoing routine clinical care for RRMS in MENA Region

DETAILED DESCRIPTION:
This is an observational, multi-center, prospective, cohort study, where no visits or intervention(s) additional to the daily practice will be performed. In the study sites, patients undergoing routine clinical care for RRMS and initiated treatment with Generic DMF (Sclera® or Marovarex ®, Hikma) in accordance with the approved SPC will be followed up and assessed for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who initiate treatment with Hikma Generic DMF at baseline in accordance with the approved Summary of Product Characteristics
2. Age ≥ 18 years
3. Patients who had a diagnosis of RRMS per 2010 or 2017 revised McDonald criteria who are :

   1. Newly diagnosed who had no prior DMT, or
   2. Switched patients who had ≥1 prior DMTs, other than DMF
4. Patients who agree to participate in the study and provide a written informed consent

Exclusion Criteria:

1. Patients with previous exposure to DMF other than (Sclera® or Marovarex ®-Hikma), Fumaderm (fumaric acid esters), or compounded fumarates.
2. Patients participating in other clinical studies
3. Patients who meet any of the contraindications to the administration of the Study drug according to the approved Summary of Product Characteristics

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from different sites in Jordan, Lebanon, Algeria, Egypt and KSA
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is ARR (Annualized Relapse Rate) at 12 month. | 12 Months
  Relapses will be identified and recorded by Site investigators. A relapse is defined as any new or historical neurological symptom, not associated with fever or infection, lasting for at least 24 h and accompanied by new neurological signs. New or recurrent neurologic symptoms that occurred <30 days after the onset of a relapse as defined earlier were considered part of the same relapse.

SECONDARY OUTCOMES:
Proportion of patients with Adverse Events (AEs) and Serious Adverse Events (SAEs) (including laboratory abnormalities) | up to 12 months from Initiation of Hikma DMF
Proportion of patients with AEs and SAEs (including laboratory abnormalities) leading to treatment discontinuation will be assessed | up to 12 months from Initiation of Hikma DMF
Proportion of patients experiencing a relapse over the 12 months period from Initiation of Hikma DMF | up to 12 months from Initiation of Hikma DMF
Time to First Relapse | up to 12 months from Initiation of Hikma DMF
Proportion of patients with disability progression as measured by the EDSS over time | up to 12 months from Initiation of Hikma DMF
  Disability worsening is defined as 1.5-point increase (if baseline EDSS score was 0), 1.0-point increase (if baseline EDSS score was < 5.5) or 0.5- point increase (if baseline EDSS score was ≥ 5.5) confirmed at least 6 months apart
Change in Multiple Sclerosis Impact Scale-29 Items (MSIS-29) scores over time | up to 12 months from Initiation of Hikma DMF
  The 29-item Multiple Sclerosis Impact Scale (MSIS-29) is a patient-reported outcome measure to assess the impact of MS on day-to-day life during the past 2 weeks from a patient's perspective; it measures 20 physical items and 9 psychological items.

CONTACTS AND LOCATIONS:
Locations (6):
- Algeria (2):
  - CHU Frantz FANON, Blida
  - Nedir Mohamed Hospital, Tizi Ouzou
- Egypt (3):
  - New University Hospital, Alexandria
  - Demerdash hospital (Ain Shams University), Cairo
  - Private Clinic, Cairo
- King Abdullah University Hospital (KAUH), Ar Ramtha, Jordan